CLINICAL TRIAL: NCT05626660
Title: Comparison Between Right and Left Radial Approach in Patients Undergoing Percutaneous Coronary Procedures
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerillos Alfy Ayoub Salib, Doctor, Assiut University
Other Study IDs: Coronary procedures
Record Dates: First submitted 2022-11-03; First posted 2022-11-25 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Right Radial Group
  Interventions: Other: Coronary angiography and percutaneous coronary intervention
- Left Radial Group
  Interventions: Other: Coronary angiography and percutaneous coronary intervention

INTERVENTIONS:
Other: Coronary angiography and percutaneous coronary intervention — Coronary angiography and percutaneous coronary intervention via radial approach

SUMMARY:
Our aim is to compare between right and left radial approach in patients undergoing percutaneous coronary procedures regarding feasibility and complications.

DETAILED DESCRIPTION:
The radial artery has progressively became the standard access site for percutaneous coronary procedures both diagnostic and interventional. The first trans-radial access for cardiovascular diagnostics dates to 1947.

In 1989, the first case series of 100 coronary angiographies performed through the radial access, demonstrating the safety and the fast mobilization of patients with the radial approach .

The main advantages of the radial approach are increased safety and comfort of the patients with reduction of bleeding complications and immediate post-procedure ambulation .with these advantages, current guidelines highly recommend radial access for coronary angiography and percutaneous coronary intervention.

Most clinical trials focused solely on the right radial approach and rarely consider the left radial approach. Indeed, the RRA has technical obstacles related to anatomy and clinical practice like increased incidence of tortuosity of the subclavian artery and radial-ulnar artery loop with the right radial approach.

Most operators use the right radial access as the left radial access increase operator discomfort during vascular access and procedure, especially in obese patients.

However, the left radial access has potential benefits for both the patient and operator. One of which is that the left radial approach is associated with lower fluoroscopy time compared with the right radial approach.

Left radial artery as well is an appropriate alternative access for coronary catheterization with less anatomical variations like tortuosity than the right radial artery Moreover, left radial access is preferred for right handed patients because of temporary post-procedural disability caused by hemostasis process in right radial artery access Also subclavian artery tortuosity is significantly more common on the right side and is an important cause of difficult, prolonged, or failed radial procedure.

ELIGIBILITY:
Inclusion Criteria:

* • All patients presented to assiut university cardiac catheterization laboratory and eligible for radial coronary procedures (either diagnostic or interventional )

Exclusion Criteria:

* • Patients with acute coronary syndrome.

  * Patients with chronic upper limb ischemia
  * Patients with AV fistula
  * Patients with severe renal impairment
  * Failure to successfully cannulate the radial artery

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing coronary angiography or elective PCI in assiut university heart hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Comparison between right and left radial approach in patients undergoing percutaneous coronary Procedures , is there is difference in tortuosity of the radial and subclavian arteries between both approaches ? | Baseline
  To compare the incidence of tortuosity in the radial and subclavian arteries between the right vs left radial approach.
  .
Comparison between right and left radial approach in patients undergoing percutaneous coronary Procedures regarding easiness of cannulation of left main coronary artery and right coronary artery tortuosity by assessing time needed for cannulation | baseline
  To compare the easiness of cannulation of left main (LM ) coronary artery and right coronary artery (RCA) via the two approaches by assessing time needed by the guiding wire and catheter to reach the ostia of either the left main coronary artery and right coronary artery .
Comparison between right and left radial approach in patients undergoing percutaneous coronary Procedures , is there is possible difference in the incidence of complications via the two approaches? | baseline
  To compare the incidence of complications e.g (bleeding , pseudoaneurysm formation ,e.t.c ) between the right and left radial approaches .
Comparison between right and left radial approach in patients undergoing percutaneous coronary Procedures regarding the incidence of crossover between right and left radial approaches and between radial and femoral approach . | baseline
  To compare the incidence of crossover between right and left radial arteries and femoral approach in case of marked radial spasm .

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daralammouri Y, Nazzal Z, Mosleh YS, Abdulhaq HK, Khayyat ZY, Hamshary YE, Azamtta M, Ghanim A, Awwad F, Majadla S, Maree M, Hamaida J, Ismail Y. Distal Radial Artery Access in comparison to Forearm Radial Artery Access for Cardiac Catheterization: A Randomized Controlled Trial (DARFORA Trial). J Interv Cardiol. 2022 Jul 15;2022:7698583. doi: 10.1155/2022/7698583. eCollection 2022. PMID 35911661
- [Background] Kiemeneij F. Left distal transradial access in the anatomical snuffbox for coronary angiography (ldTRA) and interventions (ldTRI). EuroIntervention. 2017 Sep 20;13(7):851-857. doi: 10.4244/EIJ-D-17-00079. PMID 28506941
- [Background] Lee OH, Roh JW, Im E, Cho DK, Jeong MH, Choi D, Kim Y. Feasibility and Safety of the Left Distal Radial Approach in Percutaneous Coronary Intervention for Bifurcation Lesions. J Clin Med. 2021 May 19;10(10):2204. doi: 10.3390/jcm10102204. PMID 34069701
- [Background] Klimek K, Swiatek M, Klocek K, Tworek M, Zwolski M, Milewski K, Janas A. Comparison of Safety and Efficiency between Tiger-2 Catheter with Right Radial Artery Access and Judkins Catheter with Left Radial Artery Access. J Clin Med. 2021 Sep 6;10(17):4020. doi: 10.3390/jcm10174020. PMID 34501468
- [Background] Burzotta F, Trani C, De Vita M, Crea F. A new operative classification of both anatomic vascular variants and physiopathologic conditions affecting transradial cardiovascular procedures. Int J Cardiol. 2010 Nov 5;145(1):120-2. doi: 10.1016/j.ijcard.2009.06.025. Epub 2009 Jul 17. PMID 19616324
- [Background] Dehghani P, Mohammad A, Bajaj R, Hong T, Suen CM, Sharieff W, Chisholm RJ, Kutryk MJ, Fam NP, Cheema AN. Mechanism and predictors of failed transradial approach for percutaneous coronary interventions. JACC Cardiovasc Interv. 2009 Nov;2(11):1057-64. doi: 10.1016/j.jcin.2009.07.014. PMID 19926044
- [Background] Kawamura Y, Yoshimachi F, Nakamura N, Yamamoto Y, Kudo T, Ikari Y. Impact of dedicated hemostasis device for distal radial arterial access with an adequate hemostasis protocol on radial arterial observation by ultrasound. Cardiovasc Interv Ther. 2021 Jan;36(1):104-110. doi: 10.1007/s12928-020-00656-4. Epub 2020 Mar 12. PMID 32166728
- [Background] Abdelazeem B, Abuelazm MT, Swed S, Gamal M, Atef M, Al-Zeftawy MA, Noori MA, Lutz A, Volgman AS. The efficacy of nitroglycerin to prevent radial artery spasm and occlusion during and after transradial catheterization: A systematic review and meta-analysis of randomized controlled trials. Clin Cardiol. 2022 Dec;45(12):1171-1183. doi: 10.1002/clc.23906. Epub 2022 Nov 6. PMID 36335609
- [Background] Kiemeneij F, Burzotta F, Fajadet J. Thirty years of transradial coronary interventions. EuroIntervention. 2022 May 15;18(1):19-21. doi: 10.4244/EIJ-E-22-00009. No abstract available. PMID 35570688
- [Background] RADNER S. Thoracal aortography by catheterization from the radial artery; preliminary report of a new technique. Acta Radiol (Stockh). 1948 Feb 28;29(2):178-80. doi: 10.3109/00016924809132437. No abstract available. PMID 18908938